CLINICAL TRIAL: NCT01671644
Title: Eeva™ Pregnancy Investigational Clinical Study: A Postmarket Follow-Up Study
Acronym: EPIC
Status: Completed | Type: Observational
Sponsor: Progyny, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012-AUX-005; TST-1872-p (Other: Auxogyn)
Record Dates: First submitted 2012-08-21; First posted 2012-08-23 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Infertility
Keywords: In vitro fertilization; Assisted reproductive therapy; Time-lapse image recording; Image analysis software
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Eeva Test Group: Day 3 embryo transfers that used Eeva predictions with morphology grading.
- Matched case control group: Day 3 embryo transfers using morphology grading only (from a matched concurrent control group).

SUMMARY:
The purpose of this postmarket study is to gather data to evaluate the impact of using Eeva with traditional morphology grading on clinical pregnancy rates.

DETAILED DESCRIPTION:
The purpose of this postmarket study is to gather data to evaluate the impact of using Eeva with traditional morphology grading on clinical pregnancy rates, as compared to a matched case control group that used morphology grading only to select embryos for transfer.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing fresh in vitro fertilization treatment using their own eggs or donor eggs.
* IVF cycle attempts ≤ 3.
* Egg age ≤ 40 years.
* Planned Day 3 embryo transfer.
* At least 5 normally fertilized eggs (2PN).
* All 2PN embryos must be imaged by Eeva.
* Normal uterine cavity as evaluated by standard methods.
* Fertilization using only ejaculated sperm (fresh or frozen) - no surgically removed sperm.
* Willing to comply with study protocol and procedures.
* Willing to provide written informed consent.

Exclusion Criteria:

* Planned preimplantation genetic diagnosis.
* Planned "freeze all" cycle (oocytes or embryos).
* Concurrent participation in another clinical study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing in vitro fertilization treatment who provide informed consent and plan to undergo Day 3 embryo transfer.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Rate of clinical pregnancy | 5-8 weeks gestational age
  To compare the rate of clinical pregnancy at approximately 5-8 weeks gestational age for the Day 3 embryo transfers that used Eeva predictions with morphology grading to that for Day 3 embryo transfers using morphology grading only (from a matched concurrent control group at each clinical site comprised of year 2011-2013 patients).

SECONDARY OUTCOMES:
Implantation rate (# of implanted embryos out of # of total embryos transferred) | 5-8 weeks gestational age.
Ongoing Pregnancy Rate (gestational week 10-12) | Gestational age week 10-12
Multiple pregnancy rate | Gestational weeks 5-8 and 10-12
Spontaneous miscarriage rate | Gestational age week 10-12

CONTACTS AND LOCATIONS:
Overall Officials: Shehua Shen, MD, ELD, Study Director — Progyny, Inc.
Locations (2):
- Gent University Hospital, Ghent, East Flanders, Belgium
- VU University Medical Center, Amsterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Kieslinger DC, De Gheselle S, Lambalk CB, De Sutter P, Kostelijk EH, Twisk JW, van Rijswijk J, Van den Abbeel E, Vergouw CG. Embryo selection using time-lapse analysis (Early Embryo Viability Assessment) in conjunction with standard morphology: a prospective two-center pilot study. Hum Reprod. 2016 Nov;31(11):2450-2457. doi: 10.1093/humrep/dew207. Epub 2016 Sep 12. PMID 27619774